CLINICAL TRIAL: NCT04178343
Title: Tomotherapy for Leptomeningeal Metastases: a Single Arm, Single Center, Phase II Trial
Brief Title: Tomotherapy for Leptomeningeal Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianping Xiao, Dr, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSNO-2015-MSD01
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Leptomeningeal Metastasis
Keywords: tomotherapy; leptomeningeal metastases; fractionated stereotactic radiotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Meningeal Metastases, with or without brain metastases
  Interventions: Radiation: tomotherapy

INTERVENTIONS:
Radiation: tomotherapy — 1. the prescription of tomotherapy: whole brain radiation (WBRT) with 40Gy in 20 fractions and concurrent boost of 60Gy of the leptomeningeal metastases;
  2. WBRT of 50Gy in 25 fractions, with dose limitation of hippocampus and brain stem; c.TMZ is used if necessary: concomitant TMZ: 75mg/m2 adjuvant TMZ: 150mg/ m2*5d, q28d, up to 6cycles.
  d. Some patients received intrathecal chemotherapy (MTX+AraC+Dex) based on the cytology of cerebrospinal fluid (CSF).

SUMMARY:
This clinical trial was designed to investigate the efficiency and toxicity of tomotherapy for leptomeningeal metastases.

DETAILED DESCRIPTION:
This is a single-arm, single center, phase II trial to investigate the feasibility and toxicity of tomotherapy for leptomeningeal metastases, which are defined as leptomeningeal metastases with or without brain metatstases.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of primary tumor and conformed meningeal metastases by enhanced MRI; KPS ≥60,or KPS ≥40 and the limitation of motion is simply caused by brain tumor that is adjacent to the motor function areas; Age: 18-75 years old; Adequate organ function:WBC≥4.0x109/L Neu ≥ 1.5x109/L Hemoglobin ≥ 110 g/L Platelets ≥100 x109/L Total bilirubin ≤ 1.5x ULN AST and ALT ≤ 1.5x ULN BUN and Cr: within the normal range.

Exclusion Criteria:

* Other clinically significant diseases (e.g.myocardial infarction within the past 6 months, severe arrhythmia); unable or unwilling to comply with the study protocol; patients who are anticipated in other clinical trials of meningeal metastases; pregnant patients or female patients whose HCG is positive; unsuitable to participate in study, that in the opinion of the treating physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 2 years
  the time from radiation to death

SECONDARY OUTCOMES:
local control | up to 1 year
  the time from radiation to leptomeningeal lesion recurrence
intracranial progress free survival | up to 1 year
  the time from radiation to leptomeningeal lesion recurrence and/or new brain metastases
progress free survival rate | up to 1 year
  the time from radiation to any progression
adverse event | up to 2 years
  acute and late toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Xiao, Dr, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No